CLINICAL TRIAL: NCT01230060
Title: A Prospective Multicenter Clinical Study to Evaluate the Safety and Effectiveness of a Bausch + Lomb One-Piece Hydrophobic Acrylic Intraocular Lens in Subjects Undergoing Cataract Extraction
Brief Title: One-Piece Hydrophobic Acrylic Intraocular Lens in Subjects Undergoing Cataract Extraction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 658
Record Dates: First submitted 2010-10-27; First posted 2010-10-28 (Estimated); Results first posted 2013-08-22 (Estimated); Last update posted 2013-08-22 (Estimated); Status verified 2013-08

CONDITIONS: Aphakia; Cataract
Keywords: ocular surgery; phacoemulsification
MeSH Terms: conditions — Aphakia; Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- enVista (Experimental): enVista One-Piece Hydrophobic Acrylic Intraocular Lens
  Interventions: Device: enVista

INTERVENTIONS:
Device: enVista — One-piece hydrophobic acrylic intraocular lens (IOL) implanted following cataract extraction surgery. Patients to be followed for 120-180 days following surgery.

SUMMARY:
The objective of this study is to evaluate the safety and effectiveness of the enVista® One-Piece Hydrophobic Acrylic intraocular lens (IOL), following primary implantation for the visual correction of aphakia in adults 18 years of age or older in whom the cataractous lens has been removed by an extracapsular cataract extraction method (eg, small incision phacoemulsification).

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a clinically documented diagnosis of age-related cataract that is considered amenable to treatment with standard phacoemulsification/extracapsular cataract extraction.
* Subjects must have a best corrected visual acuity (BCVA) equal to or worse than 20/40 in the study eye, with or without a glare source.
* Subjects must have a BCVA projected to be better than 20/30 after IOL implantation in the study eye.

Exclusion Criteria:

* Subjects with any anterior segment pathology for which extracapsular phacoemulsification cataract surgery would be contraindicated.
* Subjects with any other serious ocular pathology, or underlying serious medical conditions, which based on the Investigator's medical judgment, could confound the results of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2010-10; Primary Completion 2011-01 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Packer, MD,FACS, Study Director — Drs. Fine, Hoffman & Packer
Locations (1):
- Bausch & Lomb, Aliso Viejo, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 6 clinical sites in the US. Study started Aug 2010 and was completed June 2011.
Pre-assignment Details: 122 subjects underwent cataract extraction and implantation of the Bausch + Lomb Intraocular Lens (IOL) for the correction of aphakia.
Groups:
- enVista: enVista One-Piece Hydrophobic Acrylic Intraocular Lens
  enVista : One-piece hydrophobic acrylic intraocular lens (IOL) implanted following cataract extraction surgery. Patients to be followed for 120-180 days following surgery.
Period: Overall Study
Arm/Group | enVista
Started | 122
Completed | 121
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: All implanted eyes
Arm/Group | enVista
Number analyzed (Participants) | 122
Age Continuous [Mean (Standard Deviation); unit: years] | 69.0 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69
  Male | 53
Region of Enrollment [Number; unit: participants]
  United States | 122

OUTCOME MEASURES:

1. Primary Outcome: Visual Acuity
Description: Number of participants achieving best corrected visual acuity (BCVA) of 20/40 or better following cataract extraction and intraocular lens implantation.
Time Frame: 120-180 days (visit 4)
Population: All non missing implanted eyes, consistent set
Measure: Number; unit: Participants
Arm/Group | enVista
Number analyzed (Participants) | 108
Participants | 108 [96.6 to 100.0]

ADVERSE EVENTS:
Time Frame: 140-180 days
Arm/Group | enVista
Serious Adverse Events (participants affected / at risk) | 1/122
Other Adverse Events (participants affected / at risk) | 0/122
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | enVista (N=122)
Acute myeloid leukemia (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other